CLINICAL TRIAL: NCT05993104
Title: Investigating the Interplay of Left Atrial Geometry With Abnormal Propagation Patterns in Atrial Fibrillation
Brief Title: Shape vs Substrate in AF
Status: Withdrawn | Type: Observational
Why Stopped: Funder no longer operating so the study team is unable to deliver the study.
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Tim Betts MD MBChB FRCP, Associate Professor of Cardiovascular Medicine, Oxford University Hospitals NHS Trust
Other Study IDs: 16749
Record Dates: First submitted 2023-07-05; First posted 2023-08-15 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation, Persistent
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective observational: Retrospective observational arm recruiting >50 participants, utilising data already collected as part of standard clinical care.
  Interventions: Other: Statistical shape analysis
- Prospective single-arm: Prospective single-arm recruiting 20 participants undergoing AcQMap guided ablation.
  Interventions: Diagnostic Test: Intrachamber ultrasound
- Feasibility study: Feasibility study recruiting 10 participants.
  Interventions: Other: Statistical shape analysis

INTERVENTIONS:
Diagnostic Test: Intrachamber ultrasound — Ultrasound left atrial geometry collecting using AcQMap.
  Groups: Prospective single-arm
Other: Statistical shape analysis — Statistical shape analysis tools used to investigate left atrial geometry
  Groups: Feasibility study; Retrospective observational

SUMMARY:
Atrial fibrillation (AF) is an abnormal heart rhythm which originates from the top two chambers (atria) of the heart. It can cause significant symptoms and have severe consequences such as stroke.

Catheter ablation is a treatment for AF. It is minimally invasive, involving thin tubes known as catheters, being inserted through a blood vessel in the groin and passed to the heart under X-ray guidance. Once in the heart, regions of tissue believed responsible for the abnormal heart rhythm can be identified, and hot or cold energy used to create scar at these areas, preventing the abnormal rhythm.

Identifying these regions is a key challenge in making the treatment as effective as possible. The investigators believe that there may be a change in the shape of a participant's atria in these regions and as such identifying and treating areas of abnormal shape may be beneficial.

To investigate this, the study team propose three phases. The first, uses previously collected data to make a model of what is average atrial geometry in AF. Investigators will then compare individual participants' atrial geometries to this average shape to identify areas of geometric abnormality and see how these correspond to areas of abnormal electrical activity. In the second phase, investigators will collect new data on how much atrial geometry changes during catheter ablation procedures. Finally, in the third phase, investigators will investigate whether including geometric assessment in the catheter ablation procedure is feasible from a work flow perspective.

DETAILED DESCRIPTION:
This study will utilise the AcQMap system (Acutus Medical). This is a combined multi-electrode and imaging mapping system, with intra chamber ultrasound used to create a surface mesh of a participant's atrial anatomy. Noncontact charge-density mapping using AcQMap is novel, in that it allows whole chamber conduction to be analysed during AF. This is a distinct advantage over traditional contact mapping techniques, which are unable to globally map the inherently unstable and changing activation patterns occurring in AF. The system's AcQTrack software identifies patterns of localised propagation which may represent AF drivers and displays these on the surface mesh. They are classified as one of three phenomena (localised irregular activation [LIA], localised rotational activity [LRA], focal firing [FF]). AcQMap is the ideal tool for our investigation, given its ability to capture both global AF maps and geometric data. It is utilised routinely in clinical practice and there is an existing rich local dataset of previous cases.

Study Phases:

1. A retrospective observational phase recruiting >50 participants, utilising data already collected as part of standard clinical care. Investigators will use statistical shape analysis methods to create a left atrial shape model for perAF and see how individuals' left atrial geometries differ from this model. Investigators will then assess whether areas of abnormal geometry correlate with areas of abnormal electrical propagation in AF.
2. A prospective single-arm phase recruiting 20 participants undergoing AcQMap guided ablation. As previously mentioned, temporal stability is a defining characteristic of suitable ablation targets. Atrial geometry is dynamic, being related to phase of ventricular contraction and is also affected by an individual's volume status. To investigate variation in geometry, individuals in this substudy will have additional ultrasound geometries collected during their ablation procedure.
3. A feasibility study in 10 participants will assess our ability to include shape analysis as part of the procedural workflow for AF ablation utilising the AcQMap system.

ELIGIBILITY:
Inclusion Criteria:

Retrospective component:

* Participant gave consent for anonymised data being utilised for clinical research at time of procedure.
* Male or Female, aged 18 years or above.
* Previous AcQMap guided ablation for paroxysmal or persistent atrial fibrillation.

Prospective component:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with paroxysmal or persistent atrial fibrillation and planned for an AcQMap guided catheter ablation procedure.

Exclusion Criteria:

* Congenital cardiac abnormality.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with atrial fibrillation referred to a tertiary hospital (John Radcliffe, Oxford) for ablation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Regional deformation between participant left atrial geometry and SSM (study phase 1). | 1 year.
  Left atria will be partitioned into 6 segments: anterior, posterior, inferior, roof, septal and lateral. Regional deformation is defined by the mean proximity of these segments from their respective closest locations on the SSM.
Location of AF drivers defined by AcQTrack (study phase 1). | 1 year.
  Location defined using 6 segment model as described above (outcome 1).
Frequency of AF drivers defined by AcQTrack (study phase 1). | 1 year.
  Frequency of AcQTrack phenomena reported as #/s.
Regional change in AcQMap left atrial geometry during ablation procedure (study phase 2). | 2 years.
  Regional change defined using 6 segments as per outcome 1. Calculated as mean proximity of these segments during repeated geometry collection from their respective closest locations during initial geometry collection.
Completion of additional shape analysis (study phase 3). | 3 years.
Additional procedure time (study phase 3). | 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Betts, MD MBChB FRCP, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom